CLINICAL TRIAL: NCT01320969
Title: Effects of Mindfulness Practice on the Neural Circuitry of Conditioned Fear Extinction in Healthy Participants
Brief Title: Could Meditation Modulate the Neurobiology of Learning Not to Fear?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: University of Pennsylvania (Other); John Templeton Foundation (Other); Mind and Life Institute, Hadley, Massachusetts (Other)
Responsible Party: Principal Investigator, Britta Holzel, Research Fellow, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2010-P-002025
Record Dates: First submitted 2011-03-17; First posted 2011-03-23 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2012-05

CONDITIONS: Healthy Individuals; Highly Stressed
Keywords: mindfulness, fear conditioning

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindfulness-Based Stress Reduction course (Experimental): an eight week mindfulness-based stress reduction course
  Interventions: Behavioral: Mindfulness-Based Stress Reduction course
- Waitlist group (No Intervention): waitlist group

INTERVENTIONS:
Behavioral: Mindfulness-Based Stress Reduction course — an eight-week mindfulness-based stress reduction course
  Arms: Mindfulness-Based Stress Reduction course

SUMMARY:
It is well-established that the practice of mindfulness meditation leads to improvements in mental health and well-being and the cultivation of positive emotions. However, the neural mechanisms of these improvements are largely unknown. A few recent studies suggest that mindfulness meditation impacts the structure and function of the ventromedial prefrontal cortex, the hippocampus, and the amygdala. Interestingly, recent studies have shown that these regions are part of a brain circuit that is critical for the extinction of conditioned fear responses, and for the retention of fear extinction memory. Building on the overlap of these regions and on conceptual considerations, the project investigates whether mindfulness meditation could influence one's capacity to retain the memory of fear extinction. Meditation-naïve participants will be randomized to either a mindfulness-meditation based training or an active control training that controls for all mindfulness-unspecific components. Participants will undergo a fear conditioning, extinction and extinction recall protocol in an MRI scanner before and after the trainings. We hypothesize that participants who have practiced mindfulness meditation will show greater improvements in fear extinction memory after the course, and that these improvements will be correlated with anatomical and functional changes in the brain regions of interest. Improvements in fear extinction memory will also be related to improvements in self-reported psychological well-being. Merging the fields of an ancient spiritual tradition and a fundamental learning mechanism, the project investigates the underlying neural mechanisms of a practice for the enhancement of mental health and well-being.

ELIGIBILITY:
Inclusion Criteria:

18-65 years of age Proficient in English Right-handed Free of medication that affect cerebral metabolism Able to give informed consent High stress level (defined as a score of >= 3 on the 4-item Perceived Stress Scale).

Exclusion Criteria:

More than 10 meditation sessions of any tradition in their lifetime, or more than 5 sessions within the last year.

More than 10 yoga sessions of any tradition in their lifetime, or more than 5 sessions within the last year.

History of neurologic or psychiatric disease, substance abuse or dependence that is current or within the last year.

Major/chronic medical conditions History of head injury resulting in prolonged loss of consciousness and/or neurological sequelae History of seizures History of stroke Prior neurosurgical procedure Metal in the body, metal injury to the eyes Implanted pacemaker, medication pump, vagal stimulator, deep brain stimulator, TENS unit, or ventriculo-peritoneal shunt Pregnancy; breastfeeding or nursing Claustrophobia Weight > 350 lbs.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2010-12; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
change in MRI data | pre and post intervention or wait period; first set of MRIs within 3 weeks before the course, second set of MRIs within 3 weeks after course; MRIs will take 1.5 hours each and will occur on 2 consecutive days
  We will measure the change in functional MRI during fear conditioning, extinction, and extinction retention memory pre to post intervention. Furthermore, we will measure changes in structural MRI data, DTI data and resting state fMRI data.

SECONDARY OUTCOMES:
change in well-being | pre and post intervention or waitlist period; collected when the MRIs take place; will take about one hour each
  questionnaire data will also be collected pre and post the intervention / wait period; change in the scores will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Britta K Holzel, PhD, Principal Investigator — Massachusetts General Hospital; Mohammed R Milad, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Charlestown, Massachusetts, United States

REFERENCES:
- [Derived] Holzel BK, Brunsch V, Gard T, Greve DN, Koch K, Sorg C, Lazar SW, Milad MR. Mindfulness-Based Stress Reduction, Fear Conditioning, and The Uncinate Fasciculus: A Pilot Study. Front Behav Neurosci. 2016 Jun 15;10:124. doi: 10.3389/fnbeh.2016.00124. eCollection 2016. PMID 27378875
- See also: Related Info — http://www.posneuroscience.org/abstract-mediModu.html